CLINICAL TRIAL: NCT05124275
Title: Multicenter, Randomized, Double-Masked, Placebo-Controlled, Parallel Group Phase 2 Trial Evaluating the Safety and Efficacy of Pilocarpine Ophthalmic Topical Cream BID for the Treatment of Presbyopia
Brief Title: Safety and Efficacy of Pilocarpine Ophthalmic Topical Cream for the Treatment of Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ILUT-401-PRES
Record Dates: First submitted 2021-11-04; First posted 2021-11-17 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Presbyopia
Keywords: Pilocarpine; Refractive errors; Loss of near vision
MeSH Terms: conditions — Presbyopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pilocarpine Ophthalmic Topical Cream, Dose 1 (Experimental): Pilocarpine Ophthalmic Topical Cream, Dose 1
  Interventions: Drug: Pilocarpine Ophthalmic Topical Cream, Dose 1
- Pilocarpine Ophthalmic Topical Cream, Dose 2 (Experimental): Pilocarpine Ophthalmic Topical Cream, Dose 2
  Interventions: Drug: Pilocarpine Ophthalmic Topical Cream, Dose 2
- Pilocarpine Ophthalmic Topical Cream, Dose 3 (Experimental): Pilocarpine Ophthalmic Topical Cream, Dose 3
  Interventions: Drug: Pilocarpine Ophthalmic Topical Cream, Dose 3
- Placebo Ophthalmic Topical Cream (Placebo Comparator): Placebo Ophthalmic Topical Cream
  Interventions: Drug: Placebo Ophthalmic Topical Cream

INTERVENTIONS:
Drug: Pilocarpine Ophthalmic Topical Cream, Dose 1 — Pilocarpine Ophthalmic Topical Cream, Dose 1
  Other Names: GLK-302
  Arms: Pilocarpine Ophthalmic Topical Cream, Dose 1
Drug: Pilocarpine Ophthalmic Topical Cream, Dose 2 — Pilocarpine Ophthalmic Topical Cream, Dose 2
  Other Names: GLK-302
  Arms: Pilocarpine Ophthalmic Topical Cream, Dose 2
Drug: Pilocarpine Ophthalmic Topical Cream, Dose 3 — Pilocarpine Ophthalmic Topical Cream, Dose 3
  Other Names: GLK-302
  Arms: Pilocarpine Ophthalmic Topical Cream, Dose 3
Drug: Placebo Ophthalmic Topical Cream — Placebo Ophthalmic Topical Cream
  Other Names: Placebo
  Arms: Placebo Ophthalmic Topical Cream

SUMMARY:
This is a Multicenter, Randomized, Double-Masked Placebo-Controlled, Parallel Group Phase 2 Trial Evaluating the Safety and Efficacy of Pilocarpine Ophthalmic Topical Cream for the Treatment of Presbyopia.

ELIGIBILITY:
Inclusion Criteria:

* Presbyopic male or female 40-55 years of age
* Willing and able to provide written informed consent on the IRB/IEC approved informed consent form

Exclusion Criteria:

* Sensitivity or known allergy to pilocarpine or any of the other excipients of the formulation
* History of eczema, dermatitis or skin sensitivity to over-the-counter personal care products
* History of, or active, iritis or uveitis in either eye
* Pre-existing retinal diseases in either eye that may pre-dispose the subjects to retinal detachment

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Binocular Distance Corrected Near Visual Acuity (DCNVA) | Day 28
  Proportion of treatment responders [subjects gaining 3 lines or more in binocular distance corrected near visual acuity (DCNVA) and not losing more than 5 letters of binocular best corrected distance visual acuity (BCDVA)] 1 hour post-dose at the Day 28 visit.

SECONDARY OUTCOMES:
Proportion of treatment responders (as defined for the primary endpoint) at 0.5, 2, 4, and 6 hours post-dose at the day 28 visit. | Day 28
  Proportion of treatment responders (as defined for the primary endpoint) at 0.5, 2, 4, and 6 hours post-dose at the day 28 visit.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Glaukos Investigator, Chandler, Arizona
  - Glaukos Investigator, Sun City, Arizona
  - Glaukos Investigator, Glendale, California
  - Glaukos Investigator, Newport Beach, California
  - Glaukos Investigator, Petaluma, California
  - Glaukos Investigator, Louisville, Kentucky
  - Glaukos Investigator, Rochester, New York
  - Glaukos Investigator, Memphis, Tennessee
  - Glaukos Investigator, Houston, Texas
  - Glaukos Investigator, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No